CLINICAL TRIAL: NCT00156728
Title: Congestive Heart Failure Atrial Arrhythmia Monitoring and Pacing (CHAMP)
Brief Title: Study to Characterize Atrial Fibrillation in CHF Patients Indicated for CRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMD 228
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-11

CONDITIONS: Congestive Heart Failure, Atrial Fibrillation
Keywords: Pacemaker artificial, congestive heart failure and atrial fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

INTERVENTIONS:
Device: Vitatron biventricular pacemaker

SUMMARY:
The purpose of the study is to characterize atrial arrhythmias in patients indicated for Cardiac Resynchronization Therapy (CRT) and to monitor changes in atrial arrhythmias while CRT is provided.

DETAILED DESCRIPTION:
The combination of congestive heart failure and atrial fibrillation is a common co morbidity, although the exact prevalence of AF in the heart failure population is still unclear. Recent studies show a prevalence of AF ranging from about 10% to 50%, although the type of AF observed and investigated in these studies is not always clearly described.

A number of mechanisms attributed to congestive heart failure may contribute to the development of AF Experimental congestive heart failure promotes sustained AF by ionic remodeling and increased interstitial fibrosis. In contrast to tachycardia-mediated AF, in congestive heart failure no shortening of atrial refractoriness occurs. Atrial tissue stress caused by congestive heart failure may also contribute to promotion of AF by inducing triggered activity, affecting atrial refractoriness properties or resulting in increased tissue mass supporting re-entry [31]. Existence of these mechanisms suggests that treatment of congestive heart failure may also influence the development and progression of AF in these patients. Conversion of chronic AF has been observed in patients with congestive heart failure treated with biventricular pacing Ventricular ionic remodeling likely underlies the increased risk for proarrhythmia in heart failure patients exposed to antiarrhythmic drugs, prolonging the action potential duration , which therefore should be avoided in patients with congestive heart failure.

The independent prognostic significance of AF in heart failure patients is still not completely clear. Results from some recent studies suggest no independent prognostic significance of AF in heart failure patients Result from other large studies on congestive heart failure suggest an independent prognostic effect of AF in patients with AF and congestive heart failure, associated with an increased risk for pump failure death and all-cause mortality a significantly reduced 1-year survival and a higher mortality among heart failure patients who developed AF A recent review with regard to the mortality in studies on congestive heart failure suggests that concomitant AF does not have an additional effect on the mortality in patients with severe heart failure, but does increase the mortality in the setting of mild-to-moderate heart failure This observation may be attributed to the fact that the atrial contribution to left ventricular filling is limited in patients with severe diastolic dysfunction, whereas the atrial contribution may still be of hemodynamic importance in mild-to-moderate heart failure

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to comply with the protocol
* Patient is willing to sign written informed consent
* Patient is expected to remain available for Follow-up visits
* Patient age is 18 years and older
* patient is on a stable medication regimen (including beta blockers) for at least 4 weeks prior to enrollment
* Baseline criteria: patients should meet all of the following criteria, to be determined at the baseline assessment procedure within 4 weeks prior to device implantation: - New York Heart Association functional classification III or IV
* QRS duration > 130 ms
* Left ventricular ejection fraction < 35% measured by echocardiography left ventricular end diastolic dimension > 55 mm measured by echocardiography

Exclusion Criteria:

* Patients with unstable angina or who have experienced an acute myocardial infarction or received coronary artery revascularization (CABG) or coronary angioplasty (PTCA) within 3 months prior to enrollment or who are candidates for CABG or PTCA
* Patients who have experienced CVA or TIA with permanent disability within 3 months prior to enrollment
* Patient on, or anticipated to require, intravenous inotropic drug therapy
* Patients with severe primary pulmonary disease (such as cor pulmonale)
* Post heart transplant patients and patients on an urgency list for cardiac transplantation
* Supine systolic blood pressure greater than 170 mm
* Patient who are not expected to survive for 8 months of study participation due to other medical conditions
* Women who are pregnant or with child bearing potential and who are not on a reliable form of birth control
* Serum creatinine greater than 250 mol/l
* Untreated hyperthyroidism
* Patients enrolled in any concurrent (drug and/or device) study
* Patients with an existing implantable cardioverter defibrillator (ICD) or indications for an ICD including those patients with sustained VT within the previous month
* Patients with permanent atrial arrhythmias. Permanent atrial arrhythmia is defined as an arrhythmia for which any possible type of cardioversion is not considered or that is recurrent within 24 hours from an attempted cardioversion
* Patients with contraindications for implantation of a cardiac pacing device
* Patients who are already implanted with a cardiac pacing device for purposes other than Cardiac Resynchronization Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172
Dates: Start 2003-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
AF burden at 6 months

SECONDARY OUTCOMES:
NYHA class,
Ejection Fraction,
all cause and sudden death,
QRS duration,
Left Ventricular End Diastolic Dimension,
QT interval and
T wave amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Bert Albers, Ms Sc PhD, Study Director — Medtronic BRC; Christophe Leclercq, MD PhD, Principal Investigator — Departement de Cardiologie et Maladies Vasculaires CHU Pontchaillou, Rennes, France
Locations (23):
- Czechia (4):
  - Fakultní Nemocnice U Sv. Anny V Brně, Brno
  - Fakultní Nemocnice S Poliklinikou Ostrava, Ostrava-Poruba
  - Institut Klinické A Experimentální Medicíny, Prague
  - Nemocnice Na Homolce, Prague
- France (12):
  - Centre Hospitalier Du Pays D'Aix, Aix-en-Provence
  - Centre Hospitalier Universitaire, Angers
  - Chru - Hôpital Cardiologique, Lille
  - Centre Hospitalier Saint Philibert, Lomme
  - Hôpital Cardiologique Louis Pradel, Lyon
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre Medico-Chirurgical Ambroise Pare, Neuilly-sur-Seine
  - Centre Hospitalier, Pau
  - Hôpital Cardiologique Du Haut-Levêque - Chu, Pessac
  - Hôpital Pontchaillou - CHU, Rennes
  - Centre Chirurgical Du Val D'Or, Saint-Cloud
  - Clinique Pasteur, Toulouse
- Ospedale Di Careggi, Florence, Italy
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - Tweesteden Ziekenhuis, Tilburg
- Klinicki Centar Srbije, Belgrade, Serbia
- Slovenský Ústav Srdcových A Cievnych Chorôb, Bratislava, Slovakia
- St. Peters Hospital, Chertsey, United Kingdom

REFERENCES:
- [Background] Remme WJ, Swedberg K; Task Force for the Diagnosis and Treatment of Chronic Heart Failure, European Society of Cardiology. Guidelines for the diagnosis and treatment of chronic heart failure. Eur Heart J. 2001 Sep;22(17):1527-60. doi: 10.1053/euhj.2001.2783. No abstract available. PMID 11492984
- [Background] Mosterd A, de Bruijne MC, Hoes AW, Deckers JW, Hofman A, Grobbee DE. Usefulness of echocardiography in detecting left ventricular dysfunction in population-based studies (The Rotterdam Study). Am J Cardiol. 1997 Jan 1;79(1):103-4. doi: 10.1016/s0002-9149(96)00691-1. PMID 9024752
- [Background] Rihal CS, Davis KB, Kennedy JW, Gersh BJ. The utility of clinical, electrocardiographic, and roentgenographic variables in the prediction of left ventricular function. Am J Cardiol. 1995 Feb 1;75(4):220-3. doi: 10.1016/0002-9149(95)80023-l. PMID 7832126
- [Background] Wheeldon NM, MacDonald TM, Flucker CJ, McKendrick AD, McDevitt DG, Struthers AD. Echocardiography in chronic heart failure in the community. Q J Med. 1993 Jan;86(1):17-23. PMID 8438044
- [Background] SOLVD Investigators; Yusuf S, Pitt B, Davis CE, Hood WB Jr, Cohn JN. Effect of enalapril on mortality and the development of heart failure in asymptomatic patients with reduced left ventricular ejection fractions. N Engl J Med. 1992 Sep 3;327(10):685-91. doi: 10.1056/NEJM199209033271003. PMID 1463530
- [Background] Kober L, Torp-Pedersen C, Carlsen JE, Bagger H, Eliasen P, Lyngborg K, Videbaek J, Cole DS, Auclert L, Pauly NC. A clinical trial of the angiotensin-converting-enzyme inhibitor trandolapril in patients with left ventricular dysfunction after myocardial infarction. Trandolapril Cardiac Evaluation (TRACE) Study Group. N Engl J Med. 1995 Dec 21;333(25):1670-6. doi: 10.1056/NEJM199512213332503. PMID 7477219
- [Background] Flather MD, Yusuf S, Kober L, Pfeffer M, Hall A, Murray G, Torp-Pedersen C, Ball S, Pogue J, Moye L, Braunwald E. Long-term ACE-inhibitor therapy in patients with heart failure or left-ventricular dysfunction: a systematic overview of data from individual patients. ACE-Inhibitor Myocardial Infarction Collaborative Group. Lancet. 2000 May 6;355(9215):1575-81. doi: 10.1016/s0140-6736(00)02212-1. PMID 10821360
- [Background] Bayliss J, Norell M, Canepa-Anson R, Sutton G, Poole-Wilson P. Untreated heart failure: clinical and neuroendocrine effects of introducing diuretics. Br Heart J. 1987 Jan;57(1):17-22. doi: 10.1136/hrt.57.1.17. PMID 3541995
- [Background] Dargie HJ. Effect of carvedilol on outcome after myocardial infarction in patients with left-ventricular dysfunction: the CAPRICORN randomised trial. Lancet. 2001 May 5;357(9266):1385-90. doi: 10.1016/s0140-6736(00)04560-8. PMID 11356434
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Khand AU, Rankin AC, Kaye GC, Cleland JG. Systematic review of the management of atrial fibrillation in patients with heart failure. Eur Heart J. 2000 Apr;21(8):614-32. doi: 10.1053/euhj.1999.1767. PMID 10731399
- [Background] Digitalis Investigation Group. The effect of digoxin on mortality and morbidity in patients with heart failure. N Engl J Med. 1997 Feb 20;336(8):525-33. doi: 10.1056/NEJM199702203360801. PMID 9036306
- [Background] Cazeau S, Ritter P, Lazarus A, Gras D, Backdach H, Mundler O, Mugica J. Multisite pacing for end-stage heart failure: early experience. Pacing Clin Electrophysiol. 1996 Nov;19(11 Pt 2):1748-57. doi: 10.1111/j.1540-8159.1996.tb03218.x. PMID 8945034
- [Background] Auricchio A, Stellbrink C, Block M, Sack S, Vogt J, Bakker P, Klein H, Kramer A, Ding J, Salo R, Tockman B, Pochet T, Spinelli J. Effect of pacing chamber and atrioventricular delay on acute systolic function of paced patients with congestive heart failure. The Pacing Therapies for Congestive Heart Failure Study Group. The Guidant Congestive Heart Failure Research Group. Circulation. 1999 Jun 15;99(23):2993-3001. doi: 10.1161/01.cir.99.23.2993. PMID 10368116
- [Background] Gras D, Mabo P, Tang T, Luttikuis O, Chatoor R, Pedersen AK, Tscheliessnigg HH, Deharo JC, Puglisi A, Silvestre J, Kimber S, Ross H, Ravazzi A, Paul V, Skehan D. Multisite pacing as a supplemental treatment of congestive heart failure: preliminary results of the Medtronic Inc. InSync Study. Pacing Clin Electrophysiol. 1998 Nov;21(11 Pt 2):2249-55. doi: 10.1111/j.1540-8159.1998.tb01162.x. PMID 9825328
- [Background] Stellbrink C, Auricchio A, Diem B, Breithardt OA, Kloss M, Schondube FA, Klein H, Messmer BJ, Hanrath P. Potential benefit of biventricular pacing in patients with congestive heart failure and ventricular tachyarrhythmia. Am J Cardiol. 1999 Mar 11;83(5B):143D-150D. doi: 10.1016/s0002-9149(98)01016-9. PMID 10089857
- [Background] Saxon LA, Boehmer JP, Hummel J, Kacet S, De Marco T, Naccarelli G, Daoud E. Biventricular pacing in patients with congestive heart failure: two prospective randomized trials. The VIGOR CHF and VENTAK CHF Investigators. Am J Cardiol. 1999 Mar 11;83(5B):120D-123D. doi: 10.1016/s0002-9149(98)01012-1. PMID 10089853
- [Background] Cazeau S, Ritter P, Bakdach S, Lazarus A, Limousin M, Henao L, Mundler O, Daubert JC, Mugica J. Four chamber pacing in dilated cardiomyopathy. Pacing Clin Electrophysiol. 1994 Nov;17(11 Pt 2):1974-9. doi: 10.1111/j.1540-8159.1994.tb03783.x. PMID 7845801
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Cazeau S, Leclercq C, Lavergne T, Walker S, Varma C, Linde C, Garrigue S, Kappenberger L, Haywood GA, Santini M, Bailleul C, Daubert JC; Multisite Stimulation in Cardiomyopathies (MUSTIC) Study Investigators. Effects of multisite biventricular pacing in patients with heart failure and intraventricular conduction delay. N Engl J Med. 2001 Mar 22;344(12):873-80. doi: 10.1056/NEJM200103223441202. PMID 11259720
- [Background] Daubert JC, Ritter P, Le Breton H, Gras D, Leclercq C, Lazarus A, Mugica J, Mabo P, Cazeau S. Permanent left ventricular pacing with transvenous leads inserted into the coronary veins. Pacing Clin Electrophysiol. 1998 Jan;21(1 Pt 2):239-45. doi: 10.1111/j.1540-8159.1998.tb01096.x. PMID 9474680
- [Background] Gurley J, Lamba S, Moulton K, Miller B, Mullin J, Hine D, MIRACLE and InSync III investigators. Does the availability of multiple left heart lead and delivery systems matter for cardiac resynchronization therapy? Eur Heart J 2002; 4:Abstr Suppl: 51
- [Background] Auricchio A, Sack S, Stellbrink C, Neuzner J, Tockman B, Hoersch W, Klein H. Transvenous left ventricular pacing using a new over the wire coronary venous lead. Pacing Clin Electrophysiol 1999; 22: 717
- [Background] Achtelik M, Bocchiardo M, Trappe HJ, Gaita F, Lozano I, Niazi I, Gold M, Yong P, Duby C; VENTAK CHF/CONTAK CD Clinical Investigation Study Group. Performance of a new steroid-eluting coronary sinus lead designed for left ventricular pacing. Pacing Clin Electrophysiol. 2000 Nov;23(11 Pt 2):1741-3. doi: 10.1111/j.1540-8159.2000.tb07009.x. PMID 11139914
- [Background] Moss AJ, Hall WJ, Cannom DS, Daubert JP, Higgins SL, Klein H, Levine JH, Saksena S, Waldo AL, Wilber D, Brown MW, Heo M. Improved survival with an implanted defibrillator in patients with coronary disease at high risk for ventricular arrhythmia. Multicenter Automatic Defibrillator Implantation Trial Investigators. N Engl J Med. 1996 Dec 26;335(26):1933-40. doi: 10.1056/NEJM199612263352601. PMID 8960472
- [Background] Buxton AE, Lee KL, Fisher JD, Josephson ME, Prystowsky EN, Hafley G. A randomized study of the prevention of sudden death in patients with coronary artery disease. Multicenter Unsustained Tachycardia Trial Investigators. N Engl J Med. 1999 Dec 16;341(25):1882-90. doi: 10.1056/NEJM199912163412503. PMID 10601507
- [Background] Salukhe TV, Francis DP, Sutton R. Comparison of medical therapy, pacing and defibrillation in heart failure (COMPANION) trial terminated early; combined biventricular pacemaker-defibrillators reduce all-cause mortality and hospitalization. Int J Cardiol. 2003 Feb;87(2-3):119-20. doi: 10.1016/s0167-5273(02)00585-5. PMID 12559527
- [Background] Walker S, Levy TM, Rex S, Brant S, Allen J, Ilsley CJ, Paul VE. Usefulness of suppression of ventricular arrhythmia by biventricular pacing in severe congestive cardiac failure. Am J Cardiol. 2000 Jul 15;86(2):231-3. doi: 10.1016/s0002-9149(00)00865-1. No abstract available. PMID 10913492
- [Background] Higgins SL, Yong P, Sheck D, McDaniel M, Bollinger F, Vadecha M, Desai S, Meyer DB. Biventricular pacing diminishes the need for implantable cardioverter defibrillator therapy. Ventak CHF Investigators. J Am Coll Cardiol. 2000 Sep;36(3):824-7. doi: 10.1016/s0735-1097(00)00795-6. PMID 10987605
- [Background] Ehrlich JR, Nattel S, Hohnloser SH. Atrial fibrillation and congestive heart failure: specific considerations at the intersection of two common and important cardiac disease sets. J Cardiovasc Electrophysiol. 2002 Apr;13(4):399-405. doi: 10.1046/j.1540-8167.2002.00399.x. PMID 12033360
- [Background] Li D, Fareh S, Leung TK, Nattel S. Promotion of atrial fibrillation by heart failure in dogs: atrial remodeling of a different sort. Circulation. 1999 Jul 6;100(1):87-95. doi: 10.1161/01.cir.100.1.87. PMID 10393686
- [Background] Leclercq C, Walker S, Linde C, Clementy J, Marshall AJ, Ritter P, Djiane P, Mabo P, Levy T, Gadler F, Bailleul C, Daubert JC. Comparative effects of permanent biventricular and right-univentricular pacing in heart failure patients with chronic atrial fibrillation. Eur Heart J. 2002 Nov;23(22):1780-7. doi: 10.1053/euhj.2002.3232. PMID 12419298
- [Background] Hohnloser SH, Singh BN. Proarrhythmia with class III antiarrhythmic drugs: definition, electrophysiologic mechanisms, incidence, predisposing factors, and clinical implications. J Cardiovasc Electrophysiol. 1995 Oct;6(10 Pt 2):920-36. doi: 10.1111/j.1540-8167.1995.tb00368.x. PMID 8548113
- [Background] Carson PE, Johnson GR, Dunkman WB, Fletcher RD, Farrell L, Cohn JN. The influence of atrial fibrillation on prognosis in mild to moderate heart failure. The V-HeFT Studies. The V-HeFT VA Cooperative Studies Group. Circulation. 1993 Jun;87(6 Suppl):VI102-10. PMID 8500233
- [Background] Crijns HJ, Van den Berg MP, Van Gelder IC, Van Veldhuisen DJ. Management of atrial fibrillation in the setting of heart failure. Eur Heart J. 1997 May;18 Suppl C:C45-9. doi: 10.1093/eurheartj/18.suppl_c.45. PMID 9152675
- [Background] Mahoney P, Kimmel S, DeNofrio D, Wahl P, Loh E. Prognostic significance of atrial fibrillation in patients at a tertiary medical center referred for heart transplantation because of severe heart failure. Am J Cardiol. 1999 Jun 1;83(11):1544-7. doi: 10.1016/s0002-9149(99)00144-7. PMID 10363868
- [Background] Dries DL, Exner DV, Gersh BJ, Domanski MJ, Waclawiw MA, Stevenson LW. Atrial fibrillation is associated with an increased risk for mortality and heart failure progression in patients with asymptomatic and symptomatic left ventricular systolic dysfunction: a retrospective analysis of the SOLVD trials. Studies of Left Ventricular Dysfunction. J Am Coll Cardiol. 1998 Sep;32(3):695-703. doi: 10.1016/s0735-1097(98)00297-6. PMID 9741514
- [Background] Middlekauff HR, Stevenson WG, Stevenson LW. Prognostic significance of atrial fibrillation in advanced heart failure. A study of 390 patients. Circulation. 1991 Jul;84(1):40-8. doi: 10.1161/01.cir.84.1.40. PMID 2060110
- [Background] Opasich C, Tavazzi L, Lucci D, Gorini M, Albanese MC, Cacciatore G, Maggioni AP. Comparison of one-year outcome in women versus men with chronic congestive heart failure. Am J Cardiol. 2000 Aug 1;86(3):353-7. doi: 10.1016/s0002-9149(00)00934-6. PMID 10922453
- [Background] van den Berg MP, van Gelder IC, van Veldhuisen DJ. Impact of atrial fibrillation on mortality in patients with chronic heart failure. Eur J Heart Fail. 2002 Oct;4(5):571-5. doi: 10.1016/s1388-9842(02)00094-6. PMID 12413498
- [Background] International Committee of Medical Journal Editors. Uniform requirements for manuscripts submitted to biomedical journals. N Engl J Med. 1991 Feb 7;324(6):424-8. doi: 10.1056/NEJM199102073240624. No abstract available. PMID 1987468
- [Background] Ansalone G, Giannantoni P, Ricci R, Trambaiolo P, Laurenti A, Fedele F, Santini M. Doppler myocardial imaging in patients with heart failure receiving biventricular pacing treatment. Am Heart J. 2001 Nov;142(5):881-96. doi: 10.1067/mhj.2001.117324. PMID 11685178
- [Background] Ansalone G, Giannantoni P, Ricci R, Trambaiolo P, Fedele F, Santini M. Doppler myocardial imaging to evaluate the effectiveness of pacing sites in patients receiving biventricular pacing. J Am Coll Cardiol. 2002 Feb 6;39(3):489-99. doi: 10.1016/s0735-1097(01)01772-7. PMID 11823088
- [Background] Bax JJ, Molhoek SG, van Erven L, Voogd PJ, Somer S, Boersma E, Steendijk P, Schalij MJ, Van der Wall EE. Usefulness of myocardial tissue Doppler echocardiography to evaluate left ventricular dyssynchrony before and after biventricular pacing in patients with idiopathic dilated cardiomyopathy. Am J Cardiol. 2003 Jan 1;91(1):94-7. doi: 10.1016/s0002-9149(02)03009-6. No abstract available. PMID 12505583
- [Background] Garrigue S, Jais P, Espil G, Labeque JN, Hocini M, Shah DC, Haissaguerre M, Clementy J. Comparison of chronic biventricular pacing between epicardial and endocardial left ventricular stimulation using Doppler tissue imaging in patients with heart failure. Am J Cardiol. 2001 Oct 15;88(8):858-62. doi: 10.1016/s0002-9149(01)01892-6. PMID 11676947
- [Background] Yu CM, Chau E, Sanderson JE, Fan K, Tang MO, Fung WH, Lin H, Kong SL, Lam YM, Hill MR, Lau CP. Tissue Doppler echocardiographic evidence of reverse remodeling and improved synchronicity by simultaneously delaying regional contraction after biventricular pacing therapy in heart failure. Circulation. 2002 Jan 29;105(4):438-45. doi: 10.1161/hc0402.102623. PMID 11815425
- [Background] Adamson PB, St John Sutton MG, Plappert TJ, Abraham WT, Hilpisch KE, Hill MR. Echo-Defined Ventricular Dysynchrony predicts magnitude of response o Cardiac Resynchronization Abstract presented during AHA Scientific Session 2002.
- [Background] St John Sutton MG, Plappert TJ, Hilpisch KE, Chinchoy E. Baseline Aortic Pre-Ejection Interval (bAPEI) as a predictor of response to Cardiac Resynchronization Therapy (CRT) Abstract presented during AHA Scientific Session 2002.
- [Background] Pitzalis MV, Iacoviello M, Romito R, Massari F, Rizzon B, Luzzi G, Guida P, Andriani A, Mastropasqua F, Rizzon P. Cardiac resynchronization therapy tailored by echocardiographic evaluation of ventricular asynchrony. J Am Coll Cardiol. 2002 Nov 6;40(9):1615-22. doi: 10.1016/s0735-1097(02)02337-9. PMID 12427414